CLINICAL TRIAL: NCT06060990
Title: Determination of Copper and Other Trace Elements in Serum Samples From Patients With Biliary Tract Cancers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KME 0120-472/2022/3
Record Dates: First submitted 2023-09-13; First posted 2023-09-29 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Trace Element Deficiency
Keywords: metastatic biliary tract cancer, biomarkers, trace elements
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Trace Elements

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open-label single arm of patients with metastatic BTCs (Other): Systemic therapy:
  Identification of trace elements as novel predictive and prognostic biomarkers for response to systemic therapy in metastatic BTCs
  Interventions: Other: trace elements

INTERVENTIONS:
Other: trace elements — trace elements as biomarkers for response to systemic therapy in metastatic BTCs

SUMMARY:
The aim of the study is to determine the total concentration of selected trace elements (Cu, Zn, Fe), the proportion of free Cu and Cu bound to ceruloplasmin and the isotopic ratio of Cu65/Cu63 in blood serum samples from healthy volunteers and cancer patients using inductively coupled plasma mass spectrometry-based methods. The results will be statistically evaluated and the potential applications of the analytical methods used in cancer diagnosis and therapy will be assessed.

DETAILED DESCRIPTION:
Copper, zinc and iron (Cu, Zn and Fe) are among the trace metals that are essential for the normal functioning of the human body. They are involved in many biochemical reactions, are cofactors of enzymes, regulate important biological processes by binding to specific receptors and transcription factors. Their concentration in the organism is influenced by many factors such as gender, age, food, environmental pollution, etc. Deregulation of trace metal homeostasis, both at the cellular and tissue level, is part of the pathology of many cancers. It accelerates the transformation of normal cells into cancerous ones, and alters the inflammatory and anti-tumour response of immune cells such as macrophages). Knowledge of the role of essential trace metals in cancer is important for the development of modern pharmaceutical and nutritional approaches aimed at restoring the balance of trace elements in the body and enhancing the beneficial effects of systemic oncological therapy. At the same time, the results of modern research on the imbalance of essential trace metals point to their usefulness in cancer diagnosis and therapy. Biliary tract cancers (BTCs) are a heterogeneous group of uncommon and rare epithelial tumours. Surgery is the only potential curative treatment for BTCs, but approximately 70% of patients are diagnosed at advanced stages due to absence of specific symptoms in early stage. Tumour markers can be diagnostic, for tumour screening and early detection, prognostic or predictive for response to systemic oncological therapy. However, widely accepted biomarkers for diagnosing and dynamically monitoring the BTCs are still lacking. Currently applied tumour markers CA 19-9 and CEA, have limited diagnostic value for BTCs because they don't have high sensitivity and specificity for BTCs. Trace elements as biomarkers in oncology are new research field for detecting, diagnosing and prediction of response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years
* cytologically or histologically verified biliary tract cancer
* no prior systemic therapy and no radiation therapy for advanced, inoperable or metastatic disease
* WHO performance status 0 - 2 (ECOG criteria)
* imaging diagnosis (CT of thoracic and abdominal organs) performed within 4 weeks prior to the first administration of systemic therapy
* disease measurable by RECIST or ECOG criteria
* signed Consent to Participate in Clinical Research form

Exclusion Criteria:

* prior systemic treatment and radiation therapy for inoperable, metastatic disease
* WHO performance status > 2 (ECOG criteria)
* contraindications to immunotherapy (known immunodeficiency or active immunosuppressive therapy or active autoimmune disease requiring treatment)
* other malignancies, except cured basal cell or squamous cell carcinoma of the skin, in situ carcinoma of the cervix or other cured solid tumours without recurrence ≥ 3 years after treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Serum copper (Cu) as a predictive biomarker of the response to systemic treatment of biliary tract cancer patients | 3 years
  The concentration of copper (Cu) in blood serum samples from healthy volunteers and biliary cancer patients will be measured to identify the differences in levels and the ratio between both groups, and to identify the serum Cu levels as a predictive biomarker of response to systemic therapy biliary tract cancer patients in the correlation with radiological CT evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Martina Reberšek, MD, PhD, Principal Investigator — Institute of Oncology Ljubljana
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No